CLINICAL TRIAL: NCT06863311
Title: EXACT: Randomized Phase II Trial of Zanzalintinib (XL092) in Combination With Immunotherapy in Patients Who Progress on Adjuvant Therapy in Clear Cell RCC
Brief Title: Trial of Zanzalintinib (XL092) in Combination With Immunotherapy in Patients Who Progress on Adjuvant Therapy in Clear Cell RCC
Acronym: EXACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karie Runcie (Other)
Collaborators: Exelixis (Industry); Columbia University (Other)
Responsible Party: Sponsor-Investigator, Karie Runcie, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-GU22-595
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: XL092 (Experimental): Study treatment will be given in 28-day (4 week) cycles. Arm A treatment will consist of XL092 60 mg orally alone and will be taken once daily continuously (Day 1-Day 28). Treatment will continue until progression by RECIST 1.1, toxicity, or other reasons as appropriate.
  Interventions: Drug: XL092
- Arm B: XL092 and Nivolumab (Experimental): Study treatment will be given in 28-day (4 week) cycles. Arm B treatment will consist of XL092 60 mg plus nivolumab 480 mg intravenously. XL092 will be taken once daily continuously (Day 1-Day 28) and nivolumab will be administered every 4 weeks (Day 1). Treatment will continue until progression by RECIST 1.1, toxicity, or other reasons as appropriate.
  Interventions: Drug: XL092; Drug: Nivolumab

INTERVENTIONS:
Drug: XL092 — 100 mg orally
Drug: Nivolumab — 480 mg intravenously.
  Arms: Arm B: XL092 and Nivolumab

SUMMARY:
The study population for this Phase 2 study will include men and women ≥ 18 with confirmed renal cell carcinoma who have progressed on adjuvant anti-PD-1/PD-L1 therapy, the current standard of care. Subjects will be randomized to Arm A or Arm B. Study treatment will be given in 28-day (4 week) cycles. Arm A treatment will consist of zanzalintinib (XL092) alone and will be taken once daily continuously (Day 1-Day 28). Arm B treatment will consist of XL092 plus nivolumab. XL092 will be taken once daily continuously (Day 1-Day 28) and nivolumab will be administered every 4 weeks (Day 1). Treatment will continue until progression by RECIST 1.1, toxicity, or other reasons as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-1 within 28 days prior to registration.
4. Advanced or metastatic RCC with a clear cell component.
5. Prior treatment must have included an anti-PD-1. Subjects must have progressed on or after adjuvant anti-PD-1 therapy. A washout period of 14 days prior to study treatment initiation is required. Subjects must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline. Unresolved grade 2 or greater toxicity from prior checkpoint inhibitor therapy will exclude a subject from enrolling. Subjects that received other systemic therapy after anti-PD1 are not eligible.
6. Measurable disease per RECIST 1.1.
7. Demonstrate adequate organ function as defined below. All screening labs are to be obtained within 2 weeks prior to registration.

   * Absolute Neutrophil Count (ANC): ≥ 1500/mm3 without granulocytes colony-stimulating factor support within 2 weeks of screening laboratory collection
   * Platelet Count (PLT): ≥ 100,000/mm3; without transfusion within 2 weeks of screening laboratory sample collection.
   * Hemoglobin (Hgb): ≥ 9 g/dL
   * Serum Creatinine OR Calculated CrCl using Cockgroft Gault equation: Serum creatinine < 1.5 upper limit of normal (ULN) OR calculated Cr Clearance >40mL/min
   * Urine protein-to-creatinine ratio (UPCR): ≤1mg/mg (≤ 113.2mg/mmol) creatinine
   * Bilirubin: ≤ 1.5 × ULN (for subjects with Gilbert's disease < 3 x ULN)
   * Aspartate aminotransferase (AST): ≤ 3 × ULN
   * Alanine aminotransferase (ALT): ≤ 3 × ULN
   * Alkaline phosphatase (ALP): ≤ 3 × ULN. For subjects with documented bone metastasis ALP ≤ 5x ULN
   * International Normalized Ratio (INR): ≤ 1.5 x ULN
   * Activated Partial Thromboplastin Time (aPTT): ≤ 1.2 × ULN
8. Females of childbearing potential must have a negative urine or serum pregnancy test within 2 weeks prior to registration. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from penile-vaginal intercourse or to use an effective method(s) of contraception. Males able to father a child who are sexually active with female of childbearing potential must be willing to abstain from penile-vaginal intercourse or to use an effective method(s) of contraception.
10. Known HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial. Testing is not required at screening unless mandated by local policy.
11. Patients with known chronic hepatitis B virus (HBV) infection, must have an undetectable HBV viral load on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. Testing is not required at screening unless mandated by local policy.
12. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Prior treatment with Zanzalintinib.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days prior to study treatment initiation.
3. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 28 days prior to study treatment initiation unless otherwise specified.
4. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.

4. Radiation therapy for bone metastasis within 14 days, any other radiation therapy within 28 days prior to study treatment initiation. Systemic treatment with radionuclides within 6 weeks prior to study treatment initiation. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.

5. Known brain metastases or cranial epidural disease. Subjects adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 28 days prior to study treatment initiation may be eligible. NOTE: Subjects with an incidental finding of an isolated brain lesion < 1 cm in diameter may be eligible after sponsor-investigator approval if the lesion is radiographically stable for 28 days prior to study treatment initiation and does not require treatment per Investigator judgement. NOTE: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of study treatment initiation.

6. Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 14 days prior to study treatment initiation.

7. Active infection requiring systemic therapy. NOTE: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.

8. Positive TB test with active mycobacterial infection requiring systemic treatment.

9. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).

10. History of severe allergic anaphylactic reactions to study drug(s) or any of their excipients.

11. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.

12. Administration of a live, attenuated vaccine within 30 days prior to study treatment initiation.

13. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis.

14. Prior organ allograft including allogeneic stem cell transplant

15. Inability to swallow oral medications. 16. Uncontrolled major cardiovascular, pulmonary, hematologic, or psychiatric illnesses that would make the subject a poor study candidate.

17. Therapeutic doses of anticoagulants are not permitted in subjects with known brain metastases at study entry. NOTE: Subjects on therapeutic doses of LMWH or specified direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban, without known brain metastases who are on a stable dose of the anticoagulant for at least 7 days prior to randomization and without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor may be enrolled.

18. Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

• Unstable or deteriorating cardiovascular disease including but not limited to the following:

* Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, Torsades de pointes).
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
* Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 12 months before first dose.
* Prior history of myocarditis. • Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-CVA/TIA arterial thromboembolic events within 6 months before to first dose. NOTE: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and treated with anticoagulation per standard of care before first dose of study treatment. Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the sponsor-investigator.

  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
* Known gastric or esophageal varices
* Tumors invading the GI-tract from external viscera.
* Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis.
* Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is definitively managed and subject is asymptomatic.
* Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. NOTE: Complete healing of an intra-abdominal abscess must be confirmed before first dose.

  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
  * Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.
  * Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. NOTE: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following sponsor-investigator approval.

    19. Other clinically significant disorders such as:
  * Any active, known or suspected autoimmune disease. NOTE: Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
  * Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 2 weeks of first dose of study treatment. NOTE: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Transient short-term use of systemic corticosteroids for allergic conditions (eg, contrast allergy) is also allowed.
  * Malabsorption syndrome.
  * Serious non-healing wound/ulcer/bone fracture. NOTE: Non-healing wounds or ulcers are permitted if due to tumor- associated skin lesions.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of life-threatening toxicity related to prior immune therapy (eg, anti-CTLA-4, or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to recur and manageable by standard of care treatment (eg, hypothyroidism).

    20. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose. Prior laparoscopic nephrectomy within 4 weeks prior to first dose. Minor surgery (eg, simple excision, tooth extraction) within 10 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose. NOTE: Fresh tumor biopsies should be performed at least 7 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.

    21. Corrected QT interval calculated by the Fridericia formula (QTcF) > 450 ms for males or > 470 ms for females per electrocardiogram (ECG) within 14 days before first dose of study treatment. NOTE: If a single ECG shows a QTcF with an absolute value > 450 ms for males or > 470 ms for females, two additional ECGs at intervals of approximately 3 minutes must be performed within 30 minutes after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

    22. Subjects with inadequately treated adrenal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 6 months
  ORR is defined as the proportion of patients with partial response and complete response per RECIST version 1.1 criteria at any time prior to 6 months

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 2 years
  Safety and tolerability will be assessed based on the severity and frequency of treatment related Grade 3 or higher adverse events graded by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Progression Free Survival (PFS) | 2 years
  PFS is defined as the time from randomization to disease progression per RECIST 1.1 or death due to any cause (Arm B).
Overall Survival (OS) | 2 years
  OS is defined as the time from randomization to death due to any cause (Arm B)
Duration of Response (DoR) | 2 years
  DoR is defined as the time of response (PR or CR) until the time of progression per RECIST or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Karie Runcie, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York